CLINICAL TRIAL: NCT00166296
Title: Study of the Efficacy and Safety of Escitalopram for the Prevention of Depressive Episodes Induced by Peg-Interferon Alpha2a and Ribavirin in Chronic Hepatitis C Patients. Randomized, Double-Blind, Placebo-Controlled Clinical Trial
Brief Title: Efficacy and Safety of Escitalopram for Prevention of Depression Induced by Peg-Interferon in Hepatitis C Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Hoffmann-La Roche (Industry); H. Lundbeck A/S (Industry)
Responsible Party: Crisanto Diez-Quevedo, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PSQHEPGTP1; EudraCT number: 2004-002982-19
Record Dates: First submitted 2005-09-09; First posted 2005-09-14 (Estimated); Results first posted 2011-03-30 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Major Depressive Disorder; Hepatitis C, Chronic
Keywords: Major depressive disorder, chemically induced.; Peginterferon alfa-2a.; Escitalopram.; Chronic hepatitis C, psychology.; Prophylactic treatment.
MeSH Terms: conditions — Depressive Disorder, Major; Hepatitis C, Chronic | interventions — Escitalopram; Dexetimide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Escitalopram (Experimental): Escitalopram, 15 mg/day
  Interventions: Drug: Escitalopram
- Placebo pill (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Escitalopram — 15 mg/day starting 2 weeks before and 12 weeks during interferon therapy
  Other Names: Cipralex
  Arms: Escitalopram
Drug: Placebo — Placebo, 15 mg/day, starting 2 weeks before and for 12 weeks during interferon therapy.
  Arms: Placebo pill

SUMMARY:
The purpose of this study is to determine whether the use of an antidepressant (escitalopram) can prevent depressive episodes that appear during the treatment with peg-interferon and ribavirin in patients with chronic hepatitis C.

DETAILED DESCRIPTION:
Chronic hepatitis C is a prevalent condition, and the main cause of chronic liver diseases, including cirrhosis and cancer. Nowadays, interferon-alfa in combination with ribavirin is the main treatment option for this condition. In the last years, interferon molecule has been modified in order to improve tolerance into pegylated interferon.

Interferon-alfa has been associated with a high prevalence of psychiatric side effects, especially major depression (up to 25% of the cases), which is one of the main concerns about using this treatment. In fact, major depression is one of the main reasons of treatment withdrawal and treatment failure.

Major depression induced by interferon-alfa can be successfully treated with antidepressants, but we don't know if antidepressants can also prevent the development of major depression, and if this can be a safe intervention. In the literature, there is only one controlled trial about this issue, in cancer patients, and some open studies in hepatitis C.

In order to evaluate the efficacy, and safety, of an antidepressant (escitalopram) for preventing peginterferon's induced depressive episodes in patients with chronic hepatitis C, we have designed this 14-weeks placebo-controlled, double-blind, randomized clinical trial. Study interventions will be started two weeks before peginterferon + ribavirin's treatment onset.

Subjects included in the study will be patients with chronic hepatitis C who are going to be treated with peginterferon-alfa2a + ribavirin, and without mental disorders requiring active psychotropic treatment.

The main variables studied will be the appearance of a major depressive episode, following Diagnostic & Statistical Manual of Mental Disorders (DSM-IV) criteria, and the total score on the Montgomery-Asberg Depression Rating Scale, along three assessment points at 4, 8 and 12 weeks of treatment with interferon. There will also be a follow-up period of up to 6 months after treatment with interferon is completed.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic hepatitis C who are going to initiate treatment with peginterferon alfa2a + ribavirin.
* Age 18-65 years.
* Signed informed consent.
* If female, they are not in fertile period or they use barrier contraceptives.
* Patients able to understand and fill written questionnaires.

Exclusion Criteria:

* Hepatic cirrhosis or carcinoma.
* Less than 4000/mm3 leucocytes, or less than 70000/mm3 platelets.
* Hemoglobin less than 11 g/dL (females) or 12 (males).
* Any risk factor for hemolysis.
* Comorbid severe medical conditions (kidney, immune system, lung, heart, thyroid, etc).
* Baseline mental disorders that require antidepressants (depressive disorders and anxiety disorders).
* Other baseline mental disorders (delirium, substance use disorders).
* Mental disorders at any time (dementia, psychotic disorders, bipolar disorders.
* Contraindications of escitalopram (hypersensibility, diabetes, patients using serotoninergic agents, drugs that enhance the risk of bleeding, or monoamineoxidase inhibitors -MAOIs-).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2005-03; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Crisanto Diez-Quevedo, MD, Principal Investigator — Germans Trias i Pujol Hospital; Ramon Planas, MD, Principal Investigator — Germans Trias i Pujol Hospital
Locations (15):
- Spain (15):
  - Fundacion Hospital Alcorcon, Alcorcón
  - Hospital Nuestra Señora de Sonsoles, Ávila
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital del Mar, Barcelona
  - Hospital Puerta de Hierro, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario La Princesa, Madrid
  - Hospital Parc Tauli, Sabadell
  - Hospital Universitario de Salamanca, Salamanca
  - Hospital Consorci Sanitari de Terrassa, Tarrasa
  - Hospital Clínico Universitario, Valencia
  - Hospital General Universitario, Valencia
  - Hospital La Fe, Valencia
  - Hospital Miguel Servet, Zaragoza

REFERENCES:
- [Result] Diez-Quevedo C, Masnou H, Planas R, Castellvi P, Gimenez D, Morillas RM, Martin-Santos R, Navines R, Sola R, Giner P, Ardevol M, Costa J, Diago M, Pretel J. Prophylactic treatment with escitalopram of pegylated interferon alfa-2a-induced depression in hepatitis C: a 12-week, randomized, double-blind, placebo-controlled trial. J Clin Psychiatry. 2011 Apr;72(4):522-8. doi: 10.4088/JCP.09m05282blu. Epub 2010 Oct 5. PMID 21034680

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited among chronic hepatitis C patients between 18 and 65 years old, referred by general practitioners between March 2005 and July 2006 to gastroenterology outpatient units in 15 academic general hospitals in Spain, who were suitable to initiate treatment with pegylated interferonalfa-2a and ribavirin.
Groups:
- Escitalopram: Patients treated with 15 mg/day of Escitalopram since 2 weeks before starting pegylated interferon and ribavirin until week 12 of antiviral treatment
- Placebo: Patients treated with placebo since 2 weeks before starting pegylated interferon and ribavirin until week 12 of antiviral treatment
Period: Overall Study
Arm/Group | Escitalopram | Placebo
Started | 67 (Randomized patients) | 66 (Randomized patients)
ANALYZED | 66 (Patients who did receive at least the first dose of study medications, included in the analysis) | 63 (Patients who did receive at least the first dose of study medications, included in the analysis)
Completed | 60 (Patients who completed both trial medication and interferon+ribavirin treatment for 12 weeks) | 57 (Patients who completed both trial medication and interferon+ribavirin treatment for 12 weeks)
Not Completed | 7 | 9
Not completed — Withdrawal by Subject | 1 | 3
Not completed — Adverse Event | 2 | 4
Not completed — Lost to Follow-up | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Escitalopram | Placebo | Total
Number analyzed (Participants) | 67 | 66 | 133
Age, Customized [Number; unit: participants]
  Between 18 and 65 years | 67 | 66 | 133
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.7 (10.6) | 44.8 (10.8) | 45.8 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 25 | 53
  Male | 39 | 41 | 80
Region of Enrollment [Number; unit: participants]
  Spain | 67 | 66 | 133

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Developed a Major Depressive Episode According to Diagnostic & Statistical Manual of Mental Disorders, 4th Edition (DSM-IV) Criteria During the First 12 Weeks of Antiviral Treatment.
Description: At least five of the symptoms have been present during the same 1-week period: depressed mood, loss of interest or pleasure, weight or appetite changes, insomnia, agitation or retardation, fatigue, feelings of worthlessness or guilt, diminished ability to think or concentrate, recurrent thoughts of death.
  At least one of the symptoms is either depressed mood or loss of interest. Diagnoses were made by a trained psychiatrist who applied the mood disorders module from the Structured Clinical Interview for DSM-IV Axis I Disorders, non-patient edition (SCID-I/NP) at each study evaluation.
Time Frame: First three months of interferon treatment.
Population: One of 67 patients allocated to the escitalopram group and 3 of 66 in placebo did not receive the first dose of study medications. Consequently, 66 patients treated with escitalopram and 63 with placebo were included in the intention to treat analysis, with a procedure of last observation carried forward (LOCF).
Measure: Number; unit: Participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 66 | 63
Participants | 5 | 2
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Test type: Superiority or Other; p = 0.441, Fisher Exact; Odds Ratio (OR) = 0.400, 95% CI 2-sided [0.075 to 2.141]

2. Primary Outcome: Number of Participants With Sustained Hepatitis C Viral Response (Negativization of Serum Hepatitis C Virus Ribonucleic Acid).
Description: Number of participants with negativization of serum hepatitis C Virus Ribonucleic Acid (HCV RNA) 6 months after concluding antiviral therapy (sustained viral response).
  Negativization was defined as the absence of detectable levels of serum HCV RNA using a polymerase chain reaction.
Time Frame: Six months after the end of interferon treatment
Population: Patients with available data for viral response 6 months after completion of interferon treatment were compared between treatment groups.
Measure: Number; unit: Participants
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 53 | 54
Participants | 36 | 38
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: Total Score in the Montgomery-Asberg Depression Rating Scale
Description: The MADRS is a 10-item scale, clinician-administered, which is sensitive to symptom change during antidepressant treatment. It has been frequently used to measure depressive symptoms during interferon-alpha therapy and exhibits improved internal consistency in patients with co-morbid medical conditions compared with other clinician-administered questionnaires.
  Items are rated on a scale of 0-6. Scores range from 0 to 60, higher scores meaning higher levels of depression.
Time Frame: 12 weeks after interferon treatment onset
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 66 | 63
Scores on a scale | 3.82 (0.57) | 4.38 (0.63)
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Test type: Superiority or Other; p = 0.443, ANOVA

4. Secondary Outcome: Total Score in the Depression Subscale of the Hospital Anxiety and Depression Scale.
Description: The Hospital Anxiety and Depression Scale (HADS) is 14-item scale, patient-administered, that allows two independent scores of depression and anxiety. It has been specially designed to apply in patients with comorbid medical conditions as it excludes somatic or vegetative symptoms from the depression subscale.
  We present data of de depression subscale. The seven-item Depression subscale yields a score of 0-21, with higher scores meaning higher levels of depressive symptoms.
Time Frame: 12 weeks after interferon treatment onset
Measure: Mean (Standard Error); unit: Scores on a Scale
Arm/Group | Escitalopram | Placebo
Number analyzed (Participants) | 66 | 63
Scores on a Scale | 2.25 (0.34) | 2.13 (0.33)
Statistical Analysis 1: Comparison: Escitalopram vs Placebo; Test type: Superiority or Other; p = 0.930, ANOVA

ADVERSE EVENTS:
Time Frame: First three months of antiviral treatment
Arm/Group | Escitalopram | Placebo
Serious Adverse Events (participants affected / at risk) | 0/66 | 0/63
Other Adverse Events (participants affected / at risk) | 60/66 | 58/66
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Escitalopram (N=66) | Placebo (N=66)
Anemia (Blood and lymphatic system disorders) | 5 | 8/63
Anxiety (Psychiatric disorders) | 10 | 11/63
Breathing problems (Respiratory, thoracic and mediastinal disorders) | 16 | 25/63
Diarrhea (Gastrointestinal disorders) | 13 | 10/63
Dizziness (General disorders) | 9 | 3/63
Dry mouth (Gastrointestinal disorders) | 14 | 17/63
Fatigue (General disorders) | 32 | 32/63
Fever (General disorders) | 7 | 6/63
Flu-like symptoms (General disorders) | 9 | 12/63
Hair loss (Skin and subcutaneous tissue disorders) | 9 | 6/63
Headache (Nervous system disorders) | 18 | 19/63
Irritability (Psychiatric disorders) | 10 | 14/63
Leukopenia / neutropenia (Blood and lymphatic system disorders) | 7 | 4/63
Loss of appetite (Gastrointestinal disorders) | 14 | 10/63
Muscle or joint pain (Musculoskeletal and connective tissue disorders) | 22 | 32/63
Nausea or vomiting (Gastrointestinal disorders) | 23 | 21/63
Sexual dysfunction (Reproductive system and breast disorders) | 9 | 3/63
Sleep disorders (Psychiatric disorders) | 23 | 23/63

LIMITATIONS AND CAVEATS:
The low depression rate found may have underpowered the study. Selection of a much less depressive sample than in other studies. Limitation to the first 12 weeks of antiviral treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No